CLINICAL TRIAL: NCT04630015
Title: Expanded Evaluation of the Survivorship Wellness Group Program in the Context of COVID-19 and Telehealth
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 20805; NCI-2020-08530 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2020-11-13; First posted 2020-11-16 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Infection; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
Keywords: COVID-19; Cancer Survivorship
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (surveys): Patients complete surveys over 5-10 minutes at baseline (i.e. before participating in the program), and at 9 and 15 weeks follow up on the impact of COVID-19 on survivorship. Patients also complete a survey assessing how patients rate telehealth classes in the Survivorship Wellness program.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Participants will complete study specific survey

SUMMARY:
This study evaluates the effects of the Survivorship Wellness Group Program following active treatment, as well as to learn from Survivorship Wellness participants about their concerns regarding the current COVID-19 pandemic. This study may help to evaluate the impact of the survivorship program on patient well-being, provide evidence for use in grant application and publications, and ultimately inform the continued improvement of survivorship care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To examine the feasibility and acceptability of implementing an interdisciplinary goal-setting clinical group program focused on domains of physical, psychological, and spiritual wellness for survivors of cancer at University of California San Francisco (UCSF).
2. To determine preliminary efficacy of the Survivorship Wellness intervention in regards to:

   1. Increasing knowledge of and perceived confidence in execution of health behavior changes in domains of physical, emotional, and spiritual wellness for survivors of cancer.
   2. Increasing quality of life.
   3. Reducing symptoms of depression and anxiety.
   4. Increasing physical activity.
3. To assess differences in patient wellbeing and in the impact of the Survivorship Wellness program during the period of COVID-19 and telehealth classes.

OUTLINE:

Patients complete surveys over 5-10 minutes at baseline (i.e. before participating in the program), and at 9 and 15 weeks follow up on the impact of COVID-19 on survivorship. Patients also complete a survey assessing how patients rate telehealth classes in the Survivorship Wellness program.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Treated for any kind of cancer at UCSF, though finished with active treatments (defined as chemotherapy, radiation, or surgery) at time of enrollment, and without evidence of current active cancer
* Sufficient cognitive ability to participate in group activities as determined by their attending medical oncologist or surgeon

Exclusion Criteria:

* Non-English speaking
* Primary cancer treatment outside of UCSF
* Currently receiving non-maintenance therapies (chemotherapy or radiation) for active cancer
* Psychiatric illness that would affect the ability to participate in a group activity

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in the Survivorship Wellness Group Program
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in the Patient Reported Outcome Measurement Information System (PROMIS) Anxiety Short Form over time | Baseline, Week 9, and Week 15, up to 15 weeks total
  The PROMIS Anxiety Short form consists of 2 items addressing patient anxiety with item response scores ranging from 1 (never) to 5 (Always). Raw scores are converted to scaled T-scores with higher scores indicating a greater level of anxiety. Significant changes over time and trends in patient reported outcomes will be analyzed via student's T-test.
Changes in the Patient Reported Outcome Measurement Information System (PROMIS) Depression Short Form over time | Baseline, Week 9, and Week 15, up to 15 weeks total
  The PROMIS Depression Short form consists of 4 items addressing patient depression with item response scores ranging from 1 (never) to 5 (Always). Raw scores are converted to scaled T-scores with higher scores indicating a greater level of depression. Significant changes over time and trends in patient reported outcomes will be analyzed via student's T-test.
Changes in the Functional Assessment of Cancer Therapy (FACT-G) scores | Baseline, Week 9, and Week 15, up to 15 weeks total
  The FACT-G is a 27-item questionnaire designed to measure four domains of health related quality of life (HRQOL) in cancer patients with 4 domains of interest: Physical, social, emotional, and functional well-being. Each tem response score ranges from 0 (not at all) to 5 (very much). The total score is a sum of the subscale scores, with a range from 0 - 108. The higher the score, the better the HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Chesney, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No